CLINICAL TRIAL: NCT07133750
Title: A Phase II, Multicenter, Open Label, Parallel Cohort Clinical Trial to Evaluate the Efficacy and Safety of PM8002 (BNT327) in Combination With Chemotherapy in First Line MSS or MSI-L/pMMR Metastatic Colorectal Cancer
Brief Title: PM8002 (BNT327) in Combination With Chemotherapy in Patients With Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PM8002-B018C-CRC-R
Record Dates: First submitted 2025-07-30; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: CRC (Colorectal Cancer)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chemotherapy regimen 1 group - PM8002 Dose 1 + chemotherapy regimen 1 (Experimental): Subjects will be administered with PM8002 (Dose 1) plus chemotherapy regimen 1 via intravenously (IV) Q2W until progression.
  Interventions: Drug: PM8002; Drug: Chemotherapy Regimen 1
- Chemotherapy regimen 1 group - PM8002 Dose 2 + chemotherapy regimen 1 (Experimental): Subjects will be administered with PM8002 (Dose 2) plus chemotherapy regimen 1 via intravenously (IV) Q2W until progression.
  Interventions: Drug: PM8002; Drug: Chemotherapy Regimen 1
- Chemotherapy regimen 2 group - PM8002 Dose 1 + chemotherapy regimen 2 (Experimental): Subjects will be administered with PM8002 (Dose 1) plus chemotherapy regimen 2 via intravenously (IV) and oral administration (PO) Q3W until progression.
  Interventions: Drug: PM8002; Drug: Chemotherapy Regimen 2
- Chemotherapy regimen 2 group - PM8002 Dose 2 + chemotherapy regimen 2 (Experimental): Subjects will be administered with PM8002 (Dose 2) plus chemotherapy regimen 2 via intravenously (IV) and oral administration (PO) Q3W until progression.
  Interventions: Drug: PM8002; Drug: Chemotherapy Regimen 2

INTERVENTIONS:
Drug: PM8002 — IV infusion
  Other Names: BNT327
Drug: Chemotherapy Regimen 1 — IV infusion
  Arms: Chemotherapy regimen 1 group - PM8002 Dose 1 + chemotherapy regimen 1; Chemotherapy regimen 1 group - PM8002 Dose 2 + chemotherapy regimen 1
Drug: Chemotherapy Regimen 2 — Oral administration and IV infusion
  Arms: Chemotherapy regimen 2 group - PM8002 Dose 1 + chemotherapy regimen 2; Chemotherapy regimen 2 group - PM8002 Dose 2 + chemotherapy regimen 2

SUMMARY:
PM8002 (BNT327) is a bispecific antibody targeting PD-L1 and VEGF. This is a phase II trial to evaluate the efficacy and safety of PM8002 in combination with chemotherapy in first line MSS or MSI-L/pMMR metastatic colorectal cancer.

DETAILED DESCRIPTION:
A multicenter, randomized, open-label study design is used, with a planned enrollment of 40 participants, 30 in the PM8002 (BNT327)+ chemotherapy regimen 1 group and 10 in the PM8002 (BNT327)+ chemotherapy regimen 2 group. The investigators make the decision on which chemotherapy regimen to be used in the participants. After combined chemotherapy regimen is confirmed, participants will be randomized to one of two dose levels of PM8002(BNT327) plus chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed informed consent form before any trial-related processes.
2. Age ≥ 18 years male or female.
3. Histologically or cytologically confirmed metastatic colorectal cancer (stage IV, UICC/AJCC staging system) that is not suitable for or cannot be radically resected surgically.
4. Participants must not have dMMR or MSI-H.
5. No prior systemic anti-tumor therapy for metastatic colorectal cancer.
6. have adequate organ function.
7. The investigator confirms at least one measurable lesion according to RECIST v1.1. A measurable lesion located in the field of previous radiation therapy or after local treatment may be selected as a target lesion if progression is confirmed.
8. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1.

Key Exclusion Criteria:

1. Received the following treatments or medications prior to starting study treatment:

   1. Received palliative local therapy, non-specific immunomodulatory therapy, or chineses herbal therapy with an anti-tumor indication within 14 days prior to study treatment.
   2. Treatment with systemic glucocorticoids (prednisone >10 mg/day or equivalent dose of other glucocorticoids) or other immunosuppressive agents within 14 days prior to initiation of study treatment. Note: treatment with local, intraocular, intra-articular, intranasal, and inhaled glucocorticosteroids and short-term prophylactic use of glucocorticoids (e.g., to prevent allergy to contrast agent) are allowed.
2. Have a major coagulation disorder or other evidence of significant bleeding risk.
3. Adverse effects of prior antitumor therapy have not returned to a CTCAE 5.0 grade rating of ≤ grade 1
4. Have a serious non-healing wound, ulcer, or bone fracture.
5. History of abdominal fistula, gastrointestinal perforation, or abdominal abscess, history of gastrointestinal obstruction, or clinical signs of gastrointestinal obstruction within 6 months prior to initiation of study treatment.
6. Severe uncontrollable intra-abdominal inflammation that requires clinical intervention, in the judgment of the investigator.
7. Have uncontrolled hypertension or poorly controlled diabetic conditions prior to study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 2 years
  Objective response rate is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.
Occurrence and severity of TEAE (treatment emergent adverse event), TRAE（treatment related adverse event）, TESAE (treatment emergent serious adverse event）, TRSAE (treatment related serious adverse event） | From the first dose of the investigational medicinal product (IMP) to the 30-day Follow-Up Visit
  AEs are graded according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0 in the combination treatment regimen.

SECONDARY OUTCOMES:
Duration of response (DoR) | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST v1.1.
Time to response (TTR) | Up to approximately 2 years
  TTR is defined as the time from the start of the treatment to the first objective tumor response observed for patients who achieve CR or PR (based on RECIST v1.1).
Progression free survival (PFS) | Up to approximately 2 years
  Progression free survival is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).
Overall survival (OS) | Up to approximately 5 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.

OTHER OUTCOMES:
Pharmacokinetic (PK) parameters: maximum concentration | Up to 30 days after last treatment
  Maximum plasma concentration [Cmax] derived from serum concentrations of PM8002(BNT327) after study drug administration.
Pharmacokinetic (PK) parameters: minimum concentration | Up to 30 days after last treatment
  Minimum plasma concentration [Cmin] derived from serum concentrations of PM8002(BNT327) after study drug administration.
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  the incidence of ADA to PM8002
PD-L1 expression, CD8+ TIL, gene mutations | Up to approximately 2 years
  PD-L1 expression in tumor and immune cells determined by IHC (immunohistochemistry), rate of CD8+ TIL determined by IHC, gene mutation type (including KRAS/NRAS/BRAF mutation)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, PhD, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No